CLINICAL TRIAL: NCT05409599
Title: Comparison of the Effects of Vestibular Exercise and Cervical Stabilization Exercise Training on Balance and Gait in Multiple Sclerosis Patients
Brief Title: The Effects of Vestibular Exercise and Cervical Stabilization Exercise Training on Balance and Gait in MS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Director, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HakanP
Record Dates: First submitted 2022-04-08; First posted 2022-06-08 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis; Vestibular; Exercises
Keywords: Multiple Sclerosis; vestibular exercises; cervical stabilization; gait
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vestibular Exercises (Active Comparator): Cawthorne-Cooksey Exercises applied to 1st group for 3 days/week for 12 weeks
  Interventions: Other: Exercises
- Cervical Stabilization Exercises (Active Comparator): cervical stabilization Exercises applied to 1st group for 3 days/week for 12 weeks
  Interventions: Other: Exercises
- Balance Exercises (Active Comparator): classical balance Exercises applied to 1st group for 3 days/week for 12 weeks
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Exercises

SUMMARY:
The population of this research consists of individuals between the ages of 18-65 with MS disease. MS patients to be included in the study will be directed by the Neurology outpatient clinic of Sanko University Hospital. All volunteers who agreed to participate in this randomized controlled pretest-posttest design study and met the sample criteria will be included in the study.Individuals who agree to participate will be divided into three groups by simple random method and closed envelope method. Vestibular exercise training group will be formed as Group 1 and Cervical stabilization exercise training group as Group 2, control group, and Group 3 as control group.Functional reach test, tandem stand test, 25 step walking test scale form, Multiple Sclerosis Quality of Life Scale form ( MSQOL-54),Fatigue Impact Scale,Beck depression inventory, MS walking scale (msys-12), dizziness disability inventory, four step square test, timed sit and stand test

, 2 minutes walking test be performed before and after treatment,

DETAILED DESCRIPTION:
Group 1: Vestibular exercise training will be given in addition to conventional treatment (including TENS, electrical stimulation and normal joint range of motion exercises) for 12 weeks. Cawthorne-Cooksey Exercises will be given as a treatment protocol for vestibular exercise training.

Group 2 :Cervical stabilization exercise training will be given in addition to conventional treatment (including Tens, electrical stimulation and normal range of motion exercises) for 12 weeks. Cervical stabilization training improves the sense of cervical proprioception as well as strength and endurance, thereby reducing joint position sense error. Cervical stabilization exercises and training, consisting of 3 stages with increasing difficulty level, will be applied.

Group3: Classical balance exercise training will be given to the control group in addition to conventional treatment (including Tens, electrical stimulation and normal range of motion exercises) for 12 weeks. These exercises were selected among the exercises routinely used in balance rehabilitation in the literature and clinic.

Balance exercise program: walking on tiptoe and heel, walking straight and diagonally on the line, standing on a balance board, supine/prone rolling on the rehabilitation ball, pelvis control in the sagittal and frontal planes on the rehabilitation ball, prone balance on the rehabilitation ball, walking on mats of different softness , was created from side walking exercises.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed with MS
* Not having received physiotherapy-oriented treatment in the last 1 year
* not have had an attack in the last 1 month and not be in the attack period

Exclusion Criteria:

* having systemic diseases such as hypertension, heart disease, diabetes mellitus, hyperlipidemia, malignancy
* individuals whose ambulation is not independent
* Those who have undergone any surgery in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Static Balance | 12 weeks
  functional reach test
Gait speed | 12 weeks
  25-step walking test
Dizziness | 12 weeks
  dizziness disability inventory
Dinamic Balance | 12 weeks
  tandem stance test
Dinamic Balance | 12 weeks
  4 square step test
Endurance | 12 weeks
  2-minute walk test
Coordination | 12 weeks
  timed sit and stand test
Postural swing | 12 weeks
  GYKO
Walkiing difficulty | 12 Weeks
  Multiple Sclerosis Walking Scale-12 (MSYS-12)

SECONDARY OUTCOMES:
Fatigue | 12 weeks
  fatigue impact scale
Depression | 12 weeks
  beck depression inventory
MSQ54 İnventory | 12 weeks
  quality of life

CONTACTS AND LOCATIONS:
Overall Officials: hakan Polat, Study Director — Sanko University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No